CLINICAL TRIAL: NCT02032329
Title: FastFES Gait Training for Stroke Patients: Efficacy of Pre-Commercial Device
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: customKYnetics (Other)
Collaborators: University of Delaware (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S4UD; R44HD065388 (NIH)
Record Dates: First submitted 2014-01-07; First posted 2014-01-10 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2014-01

CONDITIONS: Stroke; Gait
Keywords: Functional Electrical Stimulation (FES)
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FastFES (Experimental): Single Group Study - see Intervention Description
  Interventions: Device: FastFES

INTERVENTIONS:
Device: FastFES — Fast treadmill walking supplemented with FES to ankle plantarflexor and dorsiflexor muscles, using a VFT stimulation pattern. 12 weeks of 2-3x/week. Stimulation delivered using the customKYnetics study device.

SUMMARY:
The purpose of this study is to assess efficacy of a pre-commercial device capable of activating both the ankle plantarflexor and dorsiflexor muscles using electrical stimulating during treadmill-based gait training for stroke patients.

DETAILED DESCRIPTION:
Difficulty with walking is one of the most common effects of stroke. Even after rehabilitation, a majority of stroke survivors have decreased speed, endurance, confidence, and quality of walking. Walking deficits can cause risks of falls, slow walking speed, increased effort of walking, and difficulties with activities of daily living. Restoration of walking ability can improve quality of life, and is perceived as a major goal of rehabilitation by stroke survivors. There has therefore been renewed interest in research toward developing novel gait rehabilitation treatments and improving existing treatments. FastFES is one such intervention, which improves walking post-stroke using a combination of fast treadmill training and functional electrical stimulation (FES).

Ongoing research at the University of Delaware (R01NR010786) shows that a 12-week FastFES gait rehabilitation program improves walking function, activity, and community participation in stroke survivors.

In order to facilitate implementation of the FastFES gait rehabilitation program in the clinical setting, there is a need to transition from the currently used stimulation system to a more portable stimulation system. The Study Device under evaluation is a pre-commercial prototype (developed by customKYnetics, Inc.) of a clinically viable portable electrical stimulation system that can deliver FES during gait using similar timing and parameters as are being used during FastFES gait rehabilitation training in the ongoing research.

The main goal of the efficacy study is to demonstrate clinical efficacy of the customKYnetics FastFES prototype system for improving the gait of individuals with paresis secondary to stroke. Fifteen (15) post-stroke subjects who meet the inclusion/exclusion criteria will be recruited for participation in this prospective, non-randomized, non-blinded cohort interventional study.

Training (intervention sessions) will be conducted 2-3 times per week for approximately 12 weeks for a total of 36 total sessions. Functional Electrical Stimulation (FES) to the ankle plantarflexor and dorsiflexor muscle groups will be delivered during the gait cycle using a variable frequency train (VFT) stimulation pattern. Stimulation will be coordinated to the gait cycle using data from a shoe-worn inertial sensor and proprietary real-time signal processing algorithm. Stimulation will be turned on and off in 1-minute increments during the training bouts to promote motor learning. The treadmill will be set to the patient's fastest comfortable walking speed. Each intervention session will conclude with a single overground walking session without FES.

Outcome measures assessments will be performed at the following milestones: pre-intervention, after 18 training sessions, post-intervention, and at a 12-week follow-up. This Small Business Innovation Research (SBIR) funded efficacy study will mimic the study protocol used in the R01-funded randomized controlled trial (RCT). Outcomes from the SBIR cohort will be compared to non-concurrent (e.g., historical) control groups drawn from the R01-funded RCT. The main outcomes of this study will be: 1) validation of customKYnetics' prototype system for improving gait deficits; and 2) comparison of the outcome measures of patients who trained with the customKYnetics system with those from the 'fast treadmill walking with FES' arm intervention cohort in the RCT.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-80
* Chronic stroke involving cerebral cortical regions (>6 months post stroke).
* First (single) lesion
* Ambulatory but with residual gait deficit, including those who use a cane or walker and/or demonstrate asymmetry during gait
* Able to walk for 6 minutes at their self-selected speed with no orthotic support.
* Passive ankle dorsiflexion range of motion to neutral degrees with the knee extended (i.e., able to achieve an angle of 90 degrees between the shank and the foot)
* Passive hip extension of >10 degrees
* Resting heart rate between 40-100 beats per minute
* Resting blood pressure between the range of 90/60 to 170/90

Exclusion Criteria:

* Evidence of moderate to severe chronic white matter disease on MRI
* Evidence of cerebellar stroke on MRI
* History of lower extremity joint replacement due to arthritis •Score of >1 on question 1b and >0 on question 1c on the NIH Stroke Scale
* Inability to communicate with investigators
* Neglect and hemianopia
* Unexplained dizziness in the last 6 months

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-03 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in "6-minute Walk Test (6MWT) for Distance" at 12 weeks | weeks 0 and 12
  Distance (meters) walked during the 6-minute Walk Test, a standard clinical assessment of gait will be assessed at 0 and 12 weeks. Test will be performed overground without FES. Change from baseline at 12 weeks will be computed.

CONTACTS AND LOCATIONS:
Overall Officials: Stuart A Binder-Macleod, PT, PhD, Principal Investigator — University of Delaware
Locations (1):
- University of Delaware - STAR Campus, Newark, Delaware, United States